CLINICAL TRIAL: NCT03039543
Title: The Effect of Neuromuscular Blockade During Transurethral Resection of Bladder Cancer on Surgical Condition and Recovery Profiles : A Prospective, Randomized and Controlled Trial
Brief Title: Neuromuscular Blockade During Transurethral Resection of Bladder Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: MSD Korea Ltd. (Industry)
Responsible Party: Principal Investigator, Junghee Ryu, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B-1701-378-006
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- moderate neuromuscular blockade (Active Comparator): During operation, intravenous rocuronium was used to maintain moderate (TOF count of 1 or 2). Patients in moderate neuromuscular blockade are reversed with 2 mg/kg sugammadex at a TOF count of 1 or 2.
  Interventions: Drug: Rocuronium; Drug: Sugammadex
- deep neuromuscular blockade (Experimental): During operation, intravenous rocuronium was used to maintain deep (TOF count of 0 with post-tetanic count of 2) neuromuscular blockade. Patients in the deep neuromuscular blockade are reversed with 4 mg/kg sugammadex at post-tetanic count of 2.
  Interventions: Drug: Rocuronium; Drug: Sugammadex

INTERVENTIONS:
Drug: Rocuronium — Intravenous rocuronium was used to maintain moderate (TOF count of 1 or 2) neuromuscular blockade for patients with moderate neuromuscular blockade whereas intravenous rocuronium was used to maintain deep (TOF count of 0 with post-tetanic count of 2) neuromuscular blockade for patients with deep neuromuscular blockade.
  Other Names: Esmeron
Drug: Sugammadex — Patients in moderate neuromuscular blockade are reversed with 2 mg/kg sugammadex at a TOF count of 1 or 2 and patients in the deep neuromuscular blockade are reversed with 4 mg/kg sugammadex at post-tetanic count of 2.
  Other Names: Bridion

SUMMARY:
Transurethral resection of the bladder tumor (TURB) for bladder tumor excision is the mainstream treatment. However, the beneficial effects of sugammadex after general anesthesia for TURB have not been thoroughly evaluated. Investigators hypothesized that deep NMB and the use of sugammadex as a reversal agent may be associated with better endoscopic surgical condition and recovery profile compared with moderate NMB during TURB.

This study was designed to compare patients with deep neuromuscular blockade (NMB) with moderate NMB during transurethral resection of the bladder tumor (TURB) in terms of surgical condition and postoperative recovery.

DETAILED DESCRIPTION:
Transurethral resection of the bladder tumor (TURB) is the mainstream treatment of bladder cancer. TURB may be performed under regional anesthesia or general anesthesia. During regional anesthesia for TURB, obturator nerve block should be performed to prevent adductor contraction and possible inadvertent bladder perforation. Additionally, some patients prefer not to be conscious during the surgery and patients with spinal deformity or previous spinal fusion surgery are prone to fail regional anesthesia. Therefore, general anesthesia with neuromuscular blockade (NMB) is frequently conducted for patients with TURB.

During general anesthesia for TURB, NMB is needed for intubation and optimal endoscopic surgical condition via obturator nerve block. TURB is a relatively short procedure but patients with NMB usually need sufficient time to be reversed with the conventional NMB reversal agents (anticholinesterases). Additionally, inadequate reversal from NMB may result in respiratory complication during recovery. Sugammadex, a newer reversal agent, is a selective relaxant-binding agent that allows for rapid reversal of rocuronium-induced NMB. With the introduction of sugammadex, immediate reversal of deep NMB has become possible without residual NMB.

Several previous studies evaluated the effect of NMB on surgical condition for relative short surgeries such as laparoscopic cholecystectomy or laryngeal micro-surgery. They suggested that deep NMB and reversal with sugammadex improved surgical condition without postop respiratory complications. TURB is a urological endoscopic procedure performed in a narrow bladder space but the beneficial effects of deep NMB with sugammadex reversal for TURB have not been thoroughly evaluated. We hypothesized that deep NMB and the use of sugammadex as a reversal agent may be associated with better endoscopic surgical condition compared with moderate NMB during TURB. Therefore, this study was designed to compare deep NMB with moderate NMB during TURB in terms of surgical condition and recovery profiles in patients with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years
* American Society of Anesthesiologists (ASA) physical status I and II
* scheduled to undergo elective Transurethral resection of the bladder tumor (TURB)

Exclusion Criteria:

* history of neuromuscular, renal, or hepatic disease
* a body mass index (BMI) of < 18.5 or > C 30.0 kg/m2
* treatment with drugs known to interfere with neuromuscular function

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junghee Ryu, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koo BW, Oh AY, Seo KS, Han JW, Han HS, Yoon YS. Randomized Clinical Trial of Moderate Versus Deep Neuromuscular Block for Low-Pressure Pneumoperitoneum During Laparoscopic Cholecystectomy. World J Surg. 2016 Dec;40(12):2898-2903. doi: 10.1007/s00268-016-3633-8. PMID 27405749
- [Result] Naguib M, Kopman AF, Ensor JE. Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis. Br J Anaesth. 2007 Mar;98(3):302-16. doi: 10.1093/bja/ael386. PMID 17307778
- [Result] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Started | 54 | 54
Completed | 53 | 51
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Asian
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11) | 68 (10) | 69 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 46 | 42 | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 53 | 51 | 104
operation time [Mean (Standard Deviation); unit: min] | 23 (13) | 22 (13) | 23 (13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attaining a 5 (Optimal) Surgical Condition Score
Description: 5-point surgical condition scale was evaluated as follows.
  1. Extremely poor
     * unable to work because of coughing or because of the inability to obtain a endoscopic view because of inadequate muscle relaxation. Additional neuromuscular blocking agents (NMB) must be given.
  2. Poor
     * severely hampered by inadequate muscle relaxation with continuous muscle contractions, movements, or both with the hazard of tissue damage. Additional NMB is needed.
  3. Acceptable
     * a wide endoscopic view but bladder contractions, movements, or both occur regularly causing some interference with the surgeon's work. There is the need for additional NMB to prevent deterioration.
  4. Good
     * a wide endoscopic working field with sporadic muscle contractions, movements, or both. No immediate need for additional NMB unless there is the fear of deterioration.
  5. Optimal
     * a wide endoscopic working field without any movement or contractions. No additional NMB is needed.
Time Frame: immediately following the operation, an average of 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 53 | 51
Participants | 16 | 38

2. Secondary Outcome: Incidence of Postoperative Residual Curarization
Description: the number of participant with Postoperative residual curarization (PORC, TOF ratio < 0.9 )
Time Frame: at the arrival of postoperative post-anesthesia care unit (PACU), an average of 5 minutes
Population: One patient in the moderate NMB group and 3 patients in the deep NMB group were excluded from the final analysis (1 in deep NMB group: unexpected co-operation; 1 in moderate NMB group and 2 in deep NMB group: did not maintain moderate or deep NMB)
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 53 | 51
Participants | 0 | 0

3. Secondary Outcome: Recovery Time (PACU Discharge)
Description: time needed to reach a modified Aldrete score of 9
Time Frame: During PACU stay (An average of 15 minutes)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 53 | 51
minutes | 15 (0) | 15 (0)

4. Secondary Outcome: the Incidence of Desaturation
Description: Respiratory complication such as desaturation (SpO2 < 90%) were recorded during PACU stay.
Time Frame: During PACU stay (An average of 15 minutes)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 53 | 51
Participants | 0 | 0

5. Secondary Outcome: Other Postoperative Adverse Events
Description: Pain, postoperative nausea and vomiting, dry mouth, Postoperative bladder discomfort
Time Frame: During PACU stay (An average of 15 minutes)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 53 | 51
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: During study period (induction of anesthesia-PACU stay)
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03039543/SAP_000.pdf
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03039543/Prot_001.pdf